CLINICAL TRIAL: NCT00975702
Title: Phase III Study of Efficacy of Remote Ischemic Preconditioning in Improving Outcomes in Organ Transplantation
Brief Title: Remote Ischemic Preconditioning In Abdominal Organ Transplantation
Acronym: RIPCOT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0120080212
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Kidney Disease; Liver Disease; Pancreas Disease
Keywords: Remote ischemic preconditioning; deceased organ donors; ischemia reperfusion injury; Delayed graft function; Clinical outcomes in kidney transplant recipients; Clinical outcomes in liver transplant recipients; Clinical outcomes in pancreas transplant recipients
MeSH Terms: conditions — Kidney Diseases; Liver Diseases; Pancreatic Diseases; Reperfusion Injury; Delayed Graft Function

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- No RIPC Group (No Intervention): This group is the control group or the comparator group with RIPC
- RIPC Group (Experimental): In this group deceased donors will receive Remote Ischemic Preconditioning (RIPC) by Inflation of Pneumatic Tourniquet of the lower limb prior to organ recovery.
  Interventions: Procedure: RIPC by Inflation of Pneumatic Tourniquet

INTERVENTIONS:
Procedure: RIPC by Inflation of Pneumatic Tourniquet — Pneumatic tourniquets will be placed on both lower extremities in all deceased donor subjects. In the RIPC group the tourniquets will be inflated sequentially for 10 min each followed by deflation, approximately, 30-60 min prior to aortic crossclamping and organ perfusion.
  Arms: RIPC Group

SUMMARY:
Does remote ischemic preconditioning (RIPC) induced by a brief period of occlusion of blood flow to the lower extremity prior to organ recovery in deceased donors, improve short and long term outcomes after transplantation of kidneys, livers and pancreas? To test this hypothesis deceased organ donors will be randomized to receive either RIPC or No RIPC before organ recovery. RIPC will be induced in the operating room after commencement of procurement surgery. RIPC will be induced by tourniquet-induced occlusion of blood flow to the lower extremity for 10 minutes in each side, for a total duration of 20 minutes. The remainder of the organ recovery and organ preservation will be as per standard of practice. Recovered livers, kidneys and pancreas will be transplanted into allocated recipients. Transplantation and patient management after transplantation will be as per standard of practice.

Organ-specific function and cell injury parameters will be utilized to assess the early postoperative outcomes of individual organs and recipients. Long term outcomes will be assessed by graft and recipient survival.

DETAILED DESCRIPTION:
Deceased organ donors and recipients of kidneys, livers and pancreata from the study donors comprise the study subjects.

I. DONORS

I. A. Inclusion Criteria All deceased organ donors aged > 5 years in acute care hospitals in the donor service area of the New Jersey Organ and Tissue Sharing Network (NJTO).

I.B. Exclusion criteria

1. Tissue only donors
2. Age < 5 years
3. When it is known before organ recovery that both kidneys will be leaving New JerseyIntervention: RIPC will be induced by inflation of a tourniquet around the upper thigh to 200 mm of Hg for a period of 10 minutes. After tourniquet deflation on one side, a similar procedure will be followed immediately on the opposite side. Thus, a total period of 20 minutes of lower extremity vascular occlusion will be utilized to induce RIPC. In instances of severe trauma to one lower extremity precluding tourniquet use, we will employ two cycles of 10 minutes of tourniquet occlusion in the non-traumatized lower extremity with 10 min of reperfusion in between. RIPC will be induced after commencement of procurement surgery but completed 30-45 min before circulatory arrest and initiation of organ perfusion.

   Additionally, liver biopsies (a wedge measuring 0.75 x 0.75 cm and a Tru-cut needle biopsy from the right lobe) are performed in as soon as the abdomen is opened. A wedge (1 x 0.3 cm) kidney biopsy is performed in all donors after kidney recovery but before packing the organs. All biopsies except kidney biopsies in donors aged < 50 years, are as per standard of care. The remainder of organ recovery, organ packaging and preservation are as per standard of practice. All kidneys recovered from donors classified as Extended Criteria Donors (donor age > 60 years or age 50-59 years with two of the following three criteria- cerebrovascular cause of death, a history of hypertension, terminal serum creatinine > 1.5 mg/dL) are routinely perfused ex-vivo in a pulsatile hypothermic perfusion apparatus until transplantation.

   . This may happen in a few instances either because of excellent tissue match with recipients outside New Jersey or in high risk behavior donors where all NJ kidney transplant centers have declined donor kidneys before organ recovery
4. Deceased donors in whom a decision is made not to recover both kidneys (severe kidney disease, renal failure, etc)
5. Severe trauma to both lower extremities precluding induction of RIPC

ELIGIBILITY:
Inclusion Criteria:

* All deceased organ donors aged > 5 years in acute care hospitals in the donor service area of the New Jersey Organ and Tissue Sharing Network (NJTO).

DONORS

Exclusion Criteria:

* Tissue only donors
* Age < 5 years
* When it is known before organ recovery that both kidneys will be leaving New Jersey. This may happen in a few instances either because of excellent tissue match with recipients outside New Jersey or in high risk behavior donors where all NJ kidney transplant centers have declined donor kidneys before organ recovery
* Deceased donors in whom a decision is made not to recover both kidneys (severe kidney disease, renal failure, etc)
* Severe trauma to both lower extremities precluding induction of RIPC

RECIPIENTS - KIDNEY

Inclusion Criteria:

* Patients who receive a kidney from an enrolled donor at one of the five kidney transplant centers in New Jersey, HUH, NBIMC, SBMC, RWJUH and OLMC. No kidney recipients will be enrolled at UH because UH does not perform isolated kidney transplantation.

Exclusion Criteria :

* All live donor kidney transplants performed at participating kidney transplant centers
* Recipients of deceased donor kidneys imported from outside NJTO
* Recipients of kidneys from deceased donors < 5 years of age
* Recipients of combined liver and kidney transplantation, which are performed only at UH and OLMC. The numbers of such transplants are very few per year (<5). Also, the clinical and pathophysiological issues are different from those requiring isolated kidney transplantation
* Recipients of en bloc (both kidneys together into one recipient) kidney transplantation from study donors. It is anticipated that such instances will be very few per year (<5)
* Recipients of kidneys from deceased donors not enrolled in the study due to logistical reasons.

RECIPIENTS - LIVER

Inclusion Criteria:

* All recipients of livers from deceased donors enrolled in this study and who receive their transplants at either of the two liver transplant centers in New Jersey, UH or OLMC.

Exclusion Criteria:

* Live donor recipients
* Recipients of livers imported from outside NJTO
* Recipients of deceased donor livers from donors < 5 years of age
* Recipients of livers from deceased donors not enrolled in the study due to logistical reasons

RECIPIENTS - PANCREAS

Inclusion Criteria:

* All recipients of solid organ pancreas (isolated pancreas transplant or combined kidney pancreas transplant) from deceased donors enrolled in this study and who receive their transplants at one of the four pancreas transplant centers in New Jersey, HUH, SBMC, RWJUH and OLMC. NBIMC and UH do not perform pancreas transplantation

Exclusion Criteria

* Islet cell transplant recipients
* Recipients of deceased donor whole organ pancreas imported from outside NJ
* Recipients of pancreas from deceased donors < 5 years of age
* Recipients of pancreata from deceased donors not enrolled in the study due to logistical reasons

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2009-04; Primary Completion 2010-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Organ Recovery | 1 week
  Organs Recovered and Transplanted per donor

CONTACTS AND LOCATIONS:
Overall Officials: Baburao Koneru, M.D., Principal Investigator — UMDNJ-New Jersey Medical School
Locations (1):
- University Hospital, Newark, New Jersey, United States

REFERENCES:
- [Background] Ali ZA, Callaghan CJ, Lim E, Ali AA, Nouraei SA, Akthar AM, Boyle JR, Varty K, Kharbanda RK, Dutka DP, Gaunt ME. Remote ischemic preconditioning reduces myocardial and renal injury after elective abdominal aortic aneurysm repair: a randomized controlled trial. Circulation. 2007 Sep 11;116(11 Suppl):I98-105. doi: 10.1161/circulationaha.106.679167. PMID 17846333
- [Background] Kanoria S, Jalan R, Seifalian AM, Williams R, Davidson BR. Protocols and mechanisms for remote ischemic preconditioning: a novel method for reducing ischemia reperfusion injury. Transplantation. 2007 Aug 27;84(4):445-58. doi: 10.1097/01.tp.0000228235.55419.e8. PMID 17713425
- [Background] Cheung MM, Kharbanda RK, Konstantinov IE, Shimizu M, Frndova H, Li J, Holtby HM, Cox PN, Smallhorn JF, Van Arsdell GS, Redington AN. Randomized controlled trial of the effects of remote ischemic preconditioning on children undergoing cardiac surgery: first clinical application in humans. J Am Coll Cardiol. 2006 Jun 6;47(11):2277-82. doi: 10.1016/j.jacc.2006.01.066. Epub 2006 May 15. PMID 16750696
- [Background] Hoole SP, Heck PM, Sharples L, Khan SN, Duehmke R, Densem CG, Clarke SC, Shapiro LM, Schofield PM, O'Sullivan M, Dutka DP. Cardiac Remote Ischemic Preconditioning in Coronary Stenting (CRISP Stent) Study: a prospective, randomized control trial. Circulation. 2009 Feb 17;119(6):820-7. doi: 10.1161/CIRCULATIONAHA.108.809723. Epub 2009 Feb 2. PMID 19188504
- [Background] Hausenloy DJ, Mwamure PK, Venugopal V, Harris J, Barnard M, Grundy E, Ashley E, Vichare S, Di Salvo C, Kolvekar S, Hayward M, Keogh B, MacAllister RJ, Yellon DM. Effect of remote ischaemic preconditioning on myocardial injury in patients undergoing coronary artery bypass graft surgery: a randomised controlled trial. Lancet. 2007 Aug 18;370(9587):575-9. doi: 10.1016/S0140-6736(07)61296-3. PMID 17707752